CLINICAL TRIAL: NCT05408494
Title: Engaging Men in Weight Loss With a Game-based mHealth and Neurotraining Program: A 2 x 2 Randomized Design
Brief Title: Engaging Men in Weight Loss With a Game-based mHealth and Neurotraining Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Drexel University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Evan Forman, Professor of Psychological and Brain Sciences, Drexel University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: R01DK128524 (NIH); R01DK128524 (NIH)
Record Dates: First submitted 2022-05-27; First posted 2022-06-07 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Obesity; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: Utilizing a 2 x 2 factorial design, participants will be randomized to a mobile weight loss program that includes digital self-monitoring, simplified and self-selected dietary targets program alone or to a fully-gamified version of the program, comprised of a mobile behavior change program featuring team-based competition and digital reinforcers for attainment of streaks and milestones. Participants are also randomized to receive sham or active neurotraining, which will be integrated into the program they receive.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be blind to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Non-gamified program with sham ICT (Sham Comparator): One group will be assigned to a 12-month mobile weight loss program that includes digital self-monitoring, simplified and self-selected dietary targets (to align with neurotraining and promote autonomy , and behavioral strategies with sham.
  Interventions: Behavioral: mHealth behavioral weight loss treatment
- Non-gamified program with Active ICT (Active Comparator): One group will be assigned to a 12-month mobile weight loss program that includes digital self-monitoring, simplified and self-selected dietary targets (to align with neurotraining and promote autonomy , and behavioral strategies with active neurotraining.
  Interventions: Behavioral: mHealth behavioral weight loss treatment
- Gamified program with sham ICT (Experimental): One group will receive fully-gamified version of the program with a sham.
  Interventions: Behavioral: Gamified behavioral weight loss treatment
- Gamified program with Active ICT (Experimental): One group will receive fully-gamified version of the program with active neurotraining.
  Interventions: Behavioral: Gamified behavioral weight loss treatment

INTERVENTIONS:
Behavioral: Gamified behavioral weight loss treatment — 12-month mHealth fully-gamified version of the same program, comprised of a behavior change program with digital reinforcers for attainment of streaks and milestones, and an integrated neurotraining video game
  Arms: Gamified program with Active ICT; Gamified program with sham ICT
Behavioral: mHealth behavioral weight loss treatment — a 12-month mHealth weight loss program that includes digital self-monitoring, simplified and self-selected dietary targets, physical activity and a control (sham) non-game neurotraining
  Arms: Non-gamified program with Active ICT; Non-gamified program with sham ICT

SUMMARY:
Men in the United States have an exceptionally high prevalence of overweight and obesity, i.e., 71.3%, and 42% of men are currently attempting weight loss. However, men are dramatically underrepresented in weight loss programs. Attempts to modestly adapt standard weight loss programs have seen only minimal success. Mobile applications (mHealth apps) have attractive features, but have low male enrollment and poor efficacy as conventionally delivered. A gamified mHealth program offers the possibility of engaging men and enhancing efficacy given that (1) video gaming is highly appealing to men; (2) gamification features (e.g., digital rewards for attaining "streaks" and milestones, competition) are known enhance enjoyment and motivation and facilitate desired behaviors; and (3) "neurotraining" video games featuring repetitive action mechanics, adaptive difficulty, and feedback can train inhibitory control, a basic brain capacity to inhibit intrinsically-generated approach responses that is strongly linked to body mass and the consumption of high-calorie foods. This project evaluates long-term engagement and outcomes of a professionally-designed, game-based weight loss program. As such, 228 overweight men will be randomized to: (1) a 12-month mHealth weight loss program that includes digital self-monitoring, simplified and self-selected dietary targets, physical activity and a control (sham) non-game neurotraining, or (2) a fully-gamified version of this same program, comprised of a behavior change program featuring team-based competition, digital reinforcers for attainment of streaks and milestones, and an integrated neurotraining video game. Aims include evaluating the efficacy of the gamified program in terms of weight loss, diet and physical activity at 12 months, as well as evaluating hypothesized mediators (inhibitory control and engagement), (enjoyment and compliance) and moderators (baseline frequency of video game play and implicit preferences for Inhibitory Control Training-targeted foods).

ELIGIBILITY:
Inclusion criteria:

* Individuals must be of overweight or obese BMI (25-50 kg/m)
* Individuals must be adults (aged 18-65)
* Able to engage in physical activity (defined as walking two city blocks without stopping)
* Individuals must also provide consent for the research team to contact their personal physician, if necessary, to provide clearance for the prescribed level of physical activity (i.e., walking) or to consult about rapid weight loss
* Have moderate-to-high implicit preference for high-calorie foods
* Satisfactory completion of all enrollment procedures]

Exclusion criteria:

* Medical condition (e.g., cancer, type I diabetes, renal failure), heavy alcohol use, or psychiatric condition (e.g., active substance abuse, eating disorder) that may pose a risk to the participant during intervention or cause a change in weight
* Recently began or changed the dosage of medication that can cause significant change in weight
* History of bariatric surgery
* Weight loss of ≥ 5% in the previous 3 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All participants will identify as male.
Enrollment: 228 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Baseline Weight | Assessments will be administered at month zero.
  Weight will be measured using the Fitibit Aria wireless scale, accurate to 0.2 kg. We will instruct participants to place the scale on a flat, hard surface; weigh upon waking, without clothes, after using the bathroom, require participants to confirm monthly that they are following instructions, require participants to weigh daily, remove incorrect weights, and use the average of 5 daily weights for each timepoint.
Change from Baseline Weight at 1 month | Assessment will be administered at month one.
  Weight will be measured using the Fitibit Aria wireless scale, accurate to 0.2 kg. We will instruct participants to place the scale on a flat, hard surface; weigh upon waking, without clothes, after using the bathroom, require participants to confirm monthly that they are following instructions, require participants to weigh daily, remove incorrect weights, and use the average of 5 daily weights for each timepoint.
Change from Baseline Weight at 6 months | Assessment will be administered at month sixth.
  Weight will be measured using the Fitibit Aria wireless scale, accurate to 0.2 kg. We will instruct participants to place the scale on a flat, hard surface; weigh upon waking, without clothes, after using the bathroom, require participants to confirm monthly that they are following instructions, require participants to weigh daily, remove incorrect weights, and use the average of 5 daily weights for each timepoint.
Change from Baseline Weight at 12 months | Assessment will be administered at month twelve.
  Weight will be measured using the Fitibit Aria wireless scale, accurate to 0.2 kg. We will instruct participants to place the scale on a flat, hard surface; weigh upon waking, without clothes, after using the bathroom, require participants to confirm monthly that they are following instructions, require participants to weigh daily, remove incorrect weights, and use the average of 5 daily weights for each timepoint.

SECONDARY OUTCOMES:
Caloric intake measured using the Fitbit app's built-in dietary tracking system | Assessments will be administered at months 0, 1, 6 and 12.
  Caloric intake and intake of "red" (high calorie, "unhealthy") foods will be measured using the Fitbit app's built-in dietary tracking system and accompanying food item/calorie database. Foods tracked in Fitbit will be categorized as red foods based on their energy density.
Physical activity measured in minutes of moderate to vigorous physical activity using wrist-worn activity tracker. | Assessments will be administered at months 0, 1, 6 and 12.
  Physical activity will be measured in minutes of moderate to vigorous physical activity using the Fitbit, a wrist-worn activity tracker.

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No